CLINICAL TRIAL: NCT04533945
Title: The Feasibility of Using the FreeStyle Libre Flash Glucose Monitoring System During the Transition of Care (TOC) From Inpatient to Outpatient in Persons With Type 2 Diabetes (T2D) Using Basal/Bolus Insulin
Brief Title: Feasibility of Using the CGM During TOC From in Persons With T2D Using Insulin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-0214
Record Dates: First submitted 2020-07-20; First posted 2020-09-01 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Diabetes; Type 2 Diabetes
Keywords: Continous Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- FreeStyle Libre Device (Other): Inpatients admitted to the medical-surgical units that are eligible for the trial will have the FreeStyle Libre device will be placed by the inpatient diabetes team at the discharge and glucose log will be obtained in 2 weeks followed by Hba1c in 3 months.
  Interventions: Device: FreeStyle Libre

INTERVENTIONS:
Device: FreeStyle Libre — The Freestyle Libre is a device worn on the back of the arm to measure glucose levels in the interstitial fluid. The device is applied by the patient and can be worn for 14 days, at which time it is replaced with a new device. The device does not require calibration with blood glucose testing. A scan with the receiver or a cell phone can be used to obtain glucose levels. The device does not alarm, so scanning is the only way for a patient to know if they are hypo or hyperglycemic. Studies have shown that the use of this technology can improve glycemic control as measured by Hemoglobin A1c and glucose variability in some patients. In addition, use of this technology in the outpatient setting has been associated with both improved patient satisfaction and increased glucose monitoring

SUMMARY:
Using the Libre during the TOC with persons with T2D will improve patient glucose monitoring and satisfaction, which can potentially lead to an improvement in glycemic control and hospital utilization. This study aims to assess this with inpatients using insulin.

DETAILED DESCRIPTION:
Integrating the use of the Libre during the TOC will improve patient glucose monitoring and satisfaction, which can potentially lead to an improvement in glycemic control and hospital utilization. Inpatients admitted to the medical-surgical units would be considered based on the inclusion and exclusion criteria. If the patient qualifies they would be consented to participate in the trial. In addition they would be given a script for refills. Primary outcome is change in HbA1c and secondary outcomes at baseline and 90 days include satisfaction, number of ED/inpatient visits, completion of follow-up appointment, and duration of CGM use.

ELIGIBILITY:
Inclusion Criteria:

* Persons with T2DM
* Persons on atleast 3 injections of insulin/day
* Persons whose insurance will cover the device

Exclusion Criteria:

* Persons with adhesive allergy
* Pregnant women
* Persons with CKD 4/5 or on dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (HbA1C) | 90 days
  Change in HbA1c

SECONDARY OUTCOMES:
Satisfaction with device assessed by the FreeStyle Libre Telephone Questionnaire | 90 days
  Patient satisfaction with use of FreeStyle Libre device assessed by the FreeStyle Libre Telephone Questionnaire
Number of ED/inpatient visits | 90 days
  Number of times patients experience emergency department or inpatient visits with FreeStyle Libre device
Incidence of patients that complete of follow-up appointment | 90 days
  The incidence and ratio of patients that complete a 3 month follow-up appointment after discharge with FreeStyle Libre device
Duration of CGM use | 90 days
  Patient's duration of using FreeStyle Libre device

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health North Shore University Hospital, Manhasset, New York, United States